CLINICAL TRIAL: NCT06301438
Title: Efficacy and Safety of Dalpiciclib in HR+/HER2- Advanced Breast Cancer: a Real-world Study
Brief Title: Dalpiciclib in HR+/HER2- ABC
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Other Study IDs: LY2024-022-A
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — dalpiciclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dalpiciclib: dalpiciclib oral day 1-21, every 28 days
  Interventions: Drug: dalpiciclib

INTERVENTIONS:
Drug: dalpiciclib — dalpiciclib oral day 1-21, every 28 days

SUMMARY:
To evaluate the efficacy and safety of dalpiciclib in patients with HR-positive/HER2-positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced breast cancer
* Hormone receptor-positive and human epidermal growth factor receptor 2-negative
* ECOG 0-1

Exclusion Criteria:

* Pregnant or breastfeeding
* History of immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hormone receptor-positive and human epidermal growth factor receptor 2-negative advanced breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From the date of starting dalpiciclib to the date of first documentation of progression or death (up to approximately 1 years)
  The time from the date of starting dalpiciclib to the date of disease progression as per RECIST version 1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse events | From the date of starting dalpiciclib to the end of the treatment (up to approximately 1 year)
  Adverse events during dalpiciclib treatment will be assessed according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No